CLINICAL TRIAL: NCT04189445
Title: A Phase 2 Study of Futibatinib in Patients With Specific FGFR Aberrations
Brief Title: Futibatinib in Patients With Specific FGFR Aberrations
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor made a strategic decision to terminate the study considering enrollment challenges for some of the cohorts in the trial.
Sponsor: Taiho Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAS-120-202; 2019-004084-49 (EudraCT Number)
Record Dates: First submitted 2019-12-03; First posted 2019-12-06 (Actual); Results first posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-09

CONDITIONS: Advanced or Metastatic Solid Tumor; Advanced or Metastatic Gastric or Gastroesophageal Cancer; Myeloid or Lymphoid Neoplasms (MLN)
Keywords: Futibatinib; Gastric cancer; Gastro-esophageal junction cancer; Solid tumor; Myeloid neoplasm; Lymphoid neoplasm; FGFR; Amplification; Rearrangement; TAS-120
MeSH Terms: conditions — Neoplasm Metastasis; Stomach Neoplasms | interventions — futibatinib

STUDY DESIGN:
Intervention Model Description: The study consists of independent 3 cohorts (Cohorts A, B and C) and there is no difference in the treatment regimen between the cohorts
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Futibatinib (Cohort A) (Experimental): Participants with advanced or metastatic solid tumors harboring FGFR1-4 rearrangements received futibatinib 20 mg, oral tablets, once a day on a continuous 28-day cycle up to a maximum of 841 days.
  Interventions: Drug: Futibatinib
- Futibatinib (Cohort B) (Experimental): Participants with advanced or metastatic solid gastric or GEJ cancer harboring FGFR2 amplification received futibatinib 20 mg, oral tablets, once a day on a continuous 28-day cycle up to a maximum of 297 days.
  Interventions: Drug: Futibatinib
- Futibatinib (Cohort C) (Experimental): Participants with myeloid or lymphoid neoplasm harboring FGFR1 rearrangement were to receive futibatinib 20 mg, oral tablets, once a day on a continuous 28-day cycle until disease progression, unacceptable toxicity or other treatment discontinuation criteria are met.
  Interventions: Drug: Futibatinib

INTERVENTIONS:
Drug: Futibatinib — Futibatinib tablets were dosed orally every day on a continuous 28-day cycle
  Other Names: TAS-120

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of futibatinib in patients with FGFR aberrations in 3 distinct cohorts. Patients will be enrolled into one of 3 cohorts: patients with advanced, metastatic or locally-advanced solid tumors harboring FGFR1-4 rearrangements (excluding primary brain tumors and intrahepatic cholangiocarcinoma [iCCA]); patients with gastric or gastro-esophageal junction (GEJ) cancer harboring FGFR2 amplification; and patients with myeloid or lymphoid neoplasms with FGFR1 rearrangements.

DETAILED DESCRIPTION:
Study TAS-120-202 is an open-label, multinational, 3-arm Phase 2 study evaluating the efficacy, safety, tolerability, PK, and pharmacodynamics of futibatinib in patients with FGFR aberrations. Eligible patients will be assigned to 1 of 3 treatment cohorts based on diagnosis and FGFR gene aberration status.

Patients will receive futibatinib at an oral dose of 20 mg once a day on a continuous 28-day cycle.

The study will enroll approximately:

* Cohort A: 60 patients with locally advanced, advanced, or metastatic solid tumor harboring FGFR rearrangements other than primary brain tumor or iCCA;
* Cohort B: 35 patients with locally-advanced, advanced, or metastatic gastric cancer or gastro-esophageal junction (GEJ) with FGFR2 amplification;
* Cohort C: 20 patients with myeloid or lymphoid neoplasms (MLN) with FGFR1 rearrangements

Treatment in all cohorts will continue until disease progression, unacceptable toxicity, or any other of the criteria for treatment discontinuation is met. For patients who discontinue treatment for reasons other than disease progression, tumor assessments should be continued until radiologic disease progression is documented or until initiation of subsequent new anticancer therapy (whichever occurs first).

Patients will be followed for survival every 12 weeks (±2 weeks) until survival events (deaths) have been reported for 75% of enrolled patients or the study is terminated early by the Sponsor.

Additional cohorts may be added in the future in case of new emerging efficacy data.

ELIGIBILITY:
Inclusion Criteria:

1. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
2. Known FGFR aberration status and tumor type that meet all of the criteria for 1 of the following cohorts:

   a. Cohort A

   i. Histologically-confirmed, locally-advanced, advanced, or metastatic solid tumors harboring a FGFR1-4

ii. Measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1

iii. Had disease progression/recurrence after standard treatment for their cancer

b. Cohort B

i. Histologically-confirmed, locally-advanced, advanced, or metastatic gastric or gastroesophageal junction cancer harboring a FGFR2 amplification.

ii. Measurable disease per RECIST 1.1

iii. Received at least 2 prior systemic regimens for advanced/metastatic disease

iv. Experienced disease progression/recurrence during or after the most recent prior systemic treatment for advanced/metastatic gastric cancer or GEJ cancer

c. Cohort C

i. Confirmed myeloid or lymphoid neoplasms as defined by WHO criteria with a FGFR1 rearrangement

ii. Not a candidate for hematological stem cell transplant (HSCT) or relapsed after HSCT and donor lymphocyte infusion, and progressed and not a candidate for other therapies

Exclusion Criteria:

1. History and/or current evidence of any of the following disorders:

   1. Non-tumor related alteration of the calcium-phosphorus homeostasis that is considered clinically significant in the opinion of the Investigator
   2. Ectopic mineralization/calcification including, but not limited to, soft tissue, kidneys, intestine, or myocardia and lung, considered clinically significant in the opinion of the Investigator
   3. Retinal or corneal disorder confirmed by retinal/corneal examination and considered clinically significant in the opinion of the Investigator.
2. Prior treatment with an FGFR inhibitor
3. Brain metastases that are untreated or clinically or radiologically unstable (that is, have been stable for <1 month)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2020-08-05 (Actual); Primary Completion 2024-11-11 (Actual); Study Completion 2024-11-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (61):
- United States (11):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - UCLA Medical Center, Los Angeles, California
  - Georgetown University - Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - University of Maryland, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Henry Ford Hospital, Woodhaven, Michigan
  - Mercy Clinic Oncology and Hematology - Coletta, Oklahoma City, Oklahoma
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Houston Methodist Cancer Center, Houston, Texas
  - The University of Texas M. D. Anderson Cancer Center, Houston, Texas
- Institut Jules Bordet, Brussels, Belgium
- France (8):
  - Centre Antoine Lacassagne, Nice, Alpes Maritimes
  - Centre Paul Strauss, Strasbourg, Bas Rhin
  - Centre Georges François Leclerc, Dijon, Côte-d'Or
  - Institut Bergonié, Bordeaux, Gironde
  - Hôpital Saint-Louis, Paris, Paris
  - Centre Léon Bérard, Lyon, Rhone
  - Centre Hospitalier Lyon Sud, Pierre-Bénite, Rhone
  - Institut Gustave Roussy, Villejuif, Val De Marne
- Germany (3):
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - Universitaetsklinikum Heidelberg, Heidelberg, Baden-Wurttemberg
  - Universitaetsklinikum Koeln, Cologne, North Rhine-Westphalia
- Hong Kong (2):
  - The University of Hong Kong, Hong Kong
  - Hong Kong United Oncology Centre, Jordon
- Italy (5):
  - Istituto Scientifico Romagnolo Per Lo Studio e La Cura Dei Tumori, Meldola, Forli - Cesena
  - Ospedale Sacro Cuore Don Calabria, Negrar, Verona
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - IEO Istituto Europeo di Oncologia, Milan
  - Azienda Ospedaliera Universitaria Integrata Verona (Ospedale Borgo Trento), Verona
- Japan (6):
  - Aichi Cancer Center Hospital, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa-shi, Chiba
  - NHO Shikoku Cancer Center, Matsuyama, Ehime
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Osaka University Hospital, Suita-shi, Osaka
  - National Cancer Center Hospital, Chūōku, Tokyo-To
- Netherlands (2):
  - Antoni van Leeuwenhoek, Amsterdam
  - Erasmus Medisch Centrum, Rotterdam
- Portugal (3):
  - Centro Hospitalar de Lisboa Central, E.P.E. - Hospital de Santo António dos Capuchos, Lisbon
  - Fundação Champalimaud, Lisbon
  - Centro Hospitalar do Porto, E.P.E - Hospital de Santo Antonio, Porto
- National University Cancer Institute, Singapore, Singapore
- South Korea (5):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (8):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario HM Madrid Sanchinarro, Madrid
  - Clinica Universidad de Navarra, Pamplona
  - Hospital Universitario Virgen Macarena, Seville
  - Instituto Valenciano de Oncologia IVO, Valencia
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Universitari i Politecnic La Fe, Valencia
- Sweden (2):
  - Karolinska universitetssjukhuset - Solna, Solna
  - Akademiska Sjukhuset, Uppsala
- Turkey (Türkiye) (3):
  - Acibadem Adana Hospital, Adana
  - Acibadem Maslak Hospital, Istanbul
  - Namik Kemal University, Tekirdağ
- Sarah Cannon Research Institute UK, London, Greater London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study from 05 August 2020 to 11 November 2024.
Pre-assignment Details: A total of 115 participants were enrolled in Cohort A and Cohort B to receive futibatinib; no participants were enrolled in Cohort C.
Groups:
- Futibatinib (Cohort A): Participants with advanced or metastatic solid tumors harboring fibroblast growth factor receptor (FGFR)1-4 rearrangements received futibatinib 20 milligrams (mg), oral tablets, once a day on a continuous 28-day cycle up to a maximum of 841 days.
- Futibatinib (Cohort B): Participants with advanced or metastatic solid gastric or gastro-esophageal junction (GEJ) cancer harboring FGFR2 amplification received futibatinib 20 mg, oral tablets, once a day on a continuous 28-day cycle up to a maximum of 297 days.
Period: Overall Study
Arm/Group | Futibatinib (Cohort A) | Futibatinib (Cohort B) | Futibatinib (Cohort C)
Started | 87 | 28 | 0
Completed | 0 | 0 | 0
Not Completed | 87 | 28 | 0
Not completed — Withdrawal of consent | 8 | 1 | 0
Not completed — Study Terminated by Sponsor | 25 | 3 | 0
Not completed — Death | 54 | 24 | 0

BASELINE CHARACTERISTICS:
Population: All treated population included all participants who received at least 1 dose of study drug. No participant was enrolled in Cohort C, hence no data was collected.
Groups:
- Total: Total of all reporting groups
Arm/Group | Futibatinib (Cohort A) | Futibatinib (Cohort B) | Total
Number analyzed (Participants) | 87 | 28 | 115
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.0 (12.47) | 55.6 (13.77) | 58.9 (12.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 16 | 63
  Male | 40 | 12 | 52
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Caucasian/White | 29 | 3 | 32
  Race: Black or African American | 1 | 0 | 1
  Race: Asian | 36 | 24 | 60
  Race: Other | 1 | 0 | 1
  Race: Unknown | 20 | 1 | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 3 | 1 | 4
  Ethnicity: Not Hispanic or Latino | 62 | 26 | 88
  Ethnicity: Unknown | 22 | 1 | 23

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) Based on Independent Central Review (IRC) in Cohorts A and B
Description: ORR was defined as the percentage of participants experiencing a best overall response of partial response (PR) or complete response (CR) (per Response Evaluation Criteria in Solid Tumors, RECIST version 1.1), based on IRC of radiological images. CR was defined as disappearance of all target lesions. Any pathological lymph node must have reduction in short axis to <10 millimeters (mm). PR was defined as at least a 30% decrease in the sum of diameters of the target lesions, taking as a reference the baseline sum diameters. ORR was calculated based on the best overall response recorded from the start of treatment until progressive disease or start of subsequent new anticancer treatment. Percentages were rounded off to the nearest single decimal place.
Time Frame: At the end of every 2 cycles until disease progression (Up to 31 months)
Population: All treated population included all participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Futibatinib (Cohort A) | Futibatinib (Cohort B)
Number analyzed (Participants) | 87 | 28
percentage of participants | 6.9 [2.6 to 14.4] | 17.9 [6.1 to 36.9]

2. Primary Outcome: Complete Response (CR) Rate in Cohort C
Description: CR rate was defined as the percentage of participants who achieved a CR (per response criteria for myeloid or lymphoid neoplasm) based on investigator assessment of imaging, peripheral blood, and bone marrow. CR was defined as disappearance of all target lesions. Any pathological lymph node must have reduction in short axis to <10 mm.
Time Frame: At the end of every 2 cycles until disease progression (Up to 31 months)
Population: No participants were enrolled in Cohort C, hence no data was collected.
Arm/Group | Futibatinib (Cohort C)
Number analyzed (Participants) | 0

3. Secondary Outcome: ORR Based on Investigator Assessment in Cohorts A and B
Description: ORR was defined as the percentage of participants experiencing a best overall response of PR or CR (per RECIST 1.1), based on investigator assessment. CR was defined as disappearance of all target lesions. Any pathological lymph node must have reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of the target lesions, taking as a reference the baseline sum diameters. ORR was calculated based on the best overall response recorded from the start of treatment until progressive disease or start of subsequent new anticancer treatment. Percentages were rounded off to the nearest single decimal place.
Time Frame: At the end of every 2 cycles until disease progression (Up to 31 months)
Population: All treated population included all participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Futibatinib (Cohort A) | Futibatinib (Cohort B)
Number analyzed (Participants) | 87 | 28
percentage of participants | 9.2 [4.1 to 17.3] | 10.7 [2.3 to 28.2]

4. Secondary Outcome: Duration of Response (DOR) Based on IRC in Cohorts A, B and C
Description: DOR was defined as the time from the first documentation of response (CR or PR in based on IRC) to the first documentation of objective tumor progression or death due to any cause, whichever occurs first. CR was defined as disappearance of all target lesions. Any pathological lymph node must have reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of the target lesions, taking as a reference the baseline sum diameters. DOR was estimated using the Kaplan-Meier method.
Time Frame: At the end of every 2 cycles until disease progression (Up to 31 months)
Population: All responders population included all participants who received at least 1 dose of study drug and had a response. No participants were enrolled in Cohort C, hence no data was collected. Overall number of participants analyzed is the number of participants with events.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Futibatinib (Cohort A) | Futibatinib (Cohort B) | Futibatinib (Cohort C)
Number analyzed (Participants) | 6 | 5 | 0
months | 5.6 [3.5 to NA] — The upper limit of 95% confidence interval (CI) was not estimable due to insufficient events. | 3.9 [2.1 to NA] — The upper limit of 95% CI was not estimable due to insufficient events. |

5. Secondary Outcome: DOR Based on Investigator Assessment in Cohorts A, B and C
Description: DOR was defined as the time from the first documentation of response (CR or PR in based on Investigator Assessment) to the first documentation of objective tumor progression or death due to any cause, whichever occurs first. CR was defined as disappearance of all target lesions. Any pathological lymph node must have reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of the target lesions, taking as a reference the baseline sum diameters. DOR was estimated using the Kaplan-Meier method.
Time Frame: At the end of every 2 cycles until disease progression (Up to 31 months)
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Futibatinib (Cohort A) | Futibatinib (Cohort B) | Futibatinib (Cohort C)
Number analyzed (Participants) | 8 | 3 | 0
months | 5.6 [3.0 to NA] — The upper limit of 95% CI was not estimable due to insufficient events. | 5.6 [2.0 to NA] — The upper limit of 95% CI was not estimable due to insufficient events. |

6. Secondary Outcome: Progression- Free Survival (PFS) Based on IRC in Cohorts A, B and C
Description: PFS was defined as the time from first dose of the study therapy to the date of death (any cause) or disease progression (based on IRC), whichever occurs first. The PFS was analyzed using a Kaplan-Meier method, with PFS time being censored on the date of the last disease assessment. The 95% CI for median PFS was provided using the Kaplan-Meier procedure.
Time Frame: At the end of every 2 cycles until disease progression (Up to 31 months)
Population: All treated population included all participants who received at least 1 dose of study drug. Overall number of participants analyzed are the number of participants with reported disease progression or death. No participants were enrolled in Cohort C, hence no data was collected.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Futibatinib (Cohort A) | Futibatinib (Cohort B) | Futibatinib (Cohort C)
Number analyzed (Participants) | 71 | 23 | 0
months | 1.9 [1.8 to 3.5] | 2.9 [1.8 to 3.7] |

7. Secondary Outcome: PFS Based on Investigator Review in Cohorts A, B and C
Description: PFS was defined as the time from first dose of the study therapy to the date of death (any cause) or disease progression (based on Investigator Review), whichever occurs first. The PFS was analyzed using a Kaplan-Meier method, with PFS time being censored on the date of the last disease assessment. The 95% CI for median PFS was provided using the Kaplan-Meier procedure.
Time Frame: At the end of every 2 cycles until disease progression (Up to 31 months)
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Futibatinib (Cohort A) | Futibatinib (Cohort B) | Futibatinib (Cohort C)
Number analyzed (Participants) | 71 | 25 | 0
months | 3.3 [1.9 to 3.8] | 3.3 [2.1 to 3.7] |

8. Secondary Outcome: Overall Survival (OS) in Cohorts A, B and C
Description: OS was defined as the time from the date of first dose to the death date. Participants without a documented death date were censored on the last date they were known to be alive. The OS was presented using a Kaplan-Meier estimate. The 95% CI for median OS was provided using the Kaplan-Meier procedure.
Time Frame: Up to 31 months
Population: All treated population included all participants who received at least 1 dose of study drug. Overall number of participants analyzed are the number of participants with reported death. No participants were enrolled in Cohort C, hence no data was collected.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Futibatinib (Cohort A) | Futibatinib (Cohort B) | Futibatinib (Cohort C)
Number analyzed (Participants) | 54 | 24 | 0
months | 11.1 [7.3 to 15.6] | 5.9 [3.9 to 8.9] |

9. Secondary Outcome: Disease Control Rate (DCR) Based on IRC in Cohort A and B
Description: DCR was defined as the percentage of participants experiencing a best overall response of stable disease (SD), PR, or CR (per RECIST 1.1), based on IRC. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), referencing the smallest sum diameters while on study. PD was defined as at least a 20% increase in the sum of target lesion diameters from the smallest on study (including baseline), with an absolute increase of ≥ 5 mm, or the appearance of new lesions. CR was defined as disappearance of all target lesions. Any pathological lymph node must have reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of the target lesions, taking as a reference the baseline sum diameters. Percentages were rounded off to the nearest single decimal place.
Time Frame: At the end of every 2 cycles until disease progression (Up to 31 months)
Population: All treated population included all participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Futibatinib (Cohort A) | Futibatinib (Cohort B)
Number analyzed (Participants) | 87 | 28
percentage of participants | 37.9 [27.7 to 49.0] | 50.0 [30.6 to 69.4]

10. Secondary Outcome: DCR Based on Investigator Review in Cohort A and B
Description: DCR was defined as the percentage of participants experiencing a best overall response of SD, PR, or CR (per RECIST 1.1), based on IRC. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, referencing the smallest sum diameters while on study. PD was defined as at least a 20% increase in the sum of target lesion diameters from the smallest on study (including baseline), with an absolute increase of ≥ 5 mm, or the appearance of new lesions. CR was defined as disappearance of all target lesions. Any pathological lymph node must have reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of the target lesions, taking as a reference the baseline sum diameters. Percentages were rounded off to the nearest single decimal place.
Time Frame: At the end of every 2 cycles until disease progression (Up to 31 months)
Population: All treated population included all participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Futibatinib (Cohort A) | Futibatinib (Cohort B)
Number analyzed (Participants) | 87 | 28
percentage of participants | 52.9 [41.9 to 63.7] | 64.3 [44.1 to 81.4]

11. Secondary Outcome: CR+ Complete Response With Incomplete Hematological Recovery (CRi) Rate in Cohort C
Description: CR+CRi rate was defined as the percentage of participants who achieved a CR or CRi.
Time Frame: Up to 31 months
Population: No participants were enrolled in Cohort C, hence no data was collected.
Arm/Group | Futibatinib (Cohort C)
Number analyzed (Participants) | 0

12. Secondary Outcome: Duration of CR in Cohort C
Description: Duration of CR was defined as the time from the first documentation of CR to the first documentation of recurrence or death due to any cause, whichever occurs first.
Time Frame: Up to 31 months
Population: No participants were enrolled in Cohort C, hence no data was collected.
Arm/Group | Futibatinib (Cohort C)
Number analyzed (Participants) | 0

13. Secondary Outcome: Duration of CR+CRi in Cohort C
Description: Duration of CR+CRi was defined as the time from the first documentation of CR or CRi to the first documentation of disease relapse or death due to any cause, whichever occurs first.
Time Frame: Up to 31 months
Population: No participants were enrolled in Cohort C, hence no data was collected.
Arm/Group | Futibatinib (Cohort C)
Number analyzed (Participants) | 0

14. Secondary Outcome: Complete Cytogenetic Response (CCyR) Rate in Cohort C
Description: CCyR rate was defined as the percentage of participants who achieved a CCyR.
Time Frame: Up to 31 months
Population: No participants were enrolled in Cohort C, hence no data was collected.
Arm/Group | Futibatinib (Cohort C)
Number analyzed (Participants) | 0

15. Secondary Outcome: Partial Cytogenetic Response (PCyR) Rate in Cohort C
Description: PCyR rate was defined as the percentage of participants who achieved a PCyR.
Time Frame: Up to 31 months
Population: No participants were enrolled in Cohort C, hence no data was collected.
Arm/Group | Futibatinib (Cohort C)
Number analyzed (Participants) | 0

16. Secondary Outcome: Relapse-free Survival (RFS) in Cohort C
Description: RFS was defined as the time from first documentation of CR to the date of death (any cause) or disease relapse or death due to any cause, whichever occurs first.
Time Frame: Up to 31 months
Population: No participants were enrolled in Cohort C, hence no data was collected.
Arm/Group | Futibatinib (Cohort C)
Number analyzed (Participants) | 0

17. Secondary Outcome: Event-free Survival (EFS) in Cohort C
Description: EFS was defined as the time from first dose of study therapy to treatment failure, disease relapse after CR, or participant death due to any cause, whichever occurs first.
Time Frame: Up to 31 months
Population: No participants were enrolled in Cohort C, hence no data was collected.
Arm/Group | Futibatinib (Cohort C)
Number analyzed (Participants) | 0

18. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) - Cohort A, B and C
Description: An adverse event (AE) is defined as any untoward medical occurrence in a clinical study participant and does not necessarily have a causal relationship with the study drug. A treatment-emergent AE (TEAE) is defined as an AE that is starting or worsening at the time of or after the first dose of study drug administration and within 30 days after the last dose of study drug, and does not necessarily have a causal relationship to the use of the study drug.
Time Frame: From the first dose of study drug up to 30 days after the last dose (Up to 31 months)
Population: All treated population included all participants who received at least 1 dose of study drug. No participants were enrolled in Cohort C, hence no data was collected.
Measure: Count of Participants; unit: Participants
Arm/Group | Futibatinib (Cohort A) | Futibatinib (Cohort B) | Futibatinib (Cohort C)
Number analyzed (Participants) | 87 | 28 | 0
Participants | 87 | 27 |

ADVERSE EVENTS:
Time Frame: From the first dose of study drug up to 30 days after the last dose (Up to 31 months)
Description: All treated population included all participants who received at least 1 dose of study drug. No participants were enrolled in Cohort C, hence no data was collected.
Arm/Group | Futibatinib (Cohort A) | Futibatinib (Cohort B)
All-Cause Mortality (participants affected / at risk) | 54/87 | 24/28
Serious Adverse Events (participants affected / at risk) | 23/87 | 6/28
Other Adverse Events (participants affected / at risk) | 86/87 | 27/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Futibatinib (Cohort A) (N=87) | Futibatinib (Cohort B) (N=28)
Eyelid ptosis (Eye disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Subileus (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 2 | 1
Hepatic failure (Hepatobiliary disorders) | 1 | 0
COVID-19 (Infections and infestations) | 2 | 0
Device related infection (Infections and infestations) | 1 | 0
Escherichia sepsis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 1
Blood lactic acid increased (Investigations) | 1 | 0
General physical condition abnormal (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0
Calculus urinary (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2
Haemobilia (Hepatobiliary disorders) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Futibatinib (Cohort A) (N=87) | Futibatinib (Cohort B) (N=28)
Anaemia (Blood and lymphatic system disorders) | 16 | 3
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 2 | 0
Cardiac disorder (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Congenital dyskeratosis (Congenital, familial and genetic disorders) | 1 | 0
Deafness (Ear and labyrinth disorders) | 1 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Keratitis (Eye disorders) | 4 | 2
Dry eye (Eye disorders) | 3 | 2
Vision blurred (Eye disorders) | 3 | 1
Cataract (Eye disorders) | 2 | 1
Lacrimation increased (Eye disorders) | 2 | 1
Diplopia (Eye disorders) | 1 | 0
Eye discharge (Eye disorders) | 1 | 1
Eye disorder (Eye disorders) | 1 | 1
Ocular hyperaemia (Eye disorders) | 1 | 0
Trichiasis (Eye disorders) | 1 | 0
Xerophthalmia (Eye disorders) | 1 | 0
Retinal disorder (Eye disorders) | 0 | 2
Blepharitis (Eye disorders) | 0 | 1
Eye pain (Eye disorders) | 0 | 1
Meibomian gland dysfunction (Eye disorders) | 0 | 1
Serous retinal detachment (Eye disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 36 | 6
Constipation (Gastrointestinal disorders) | 28 | 3
Dry mouth (Gastrointestinal disorders) | 20 | 1
Abdominal pain (Gastrointestinal disorders) | 14 | 2
Stomatitis (Gastrointestinal disorders) | 12 | 2
Nausea (Gastrointestinal disorders) | 8 | 6
Vomiting (Gastrointestinal disorders) | 8 | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 | 1
Dyspepsia (Gastrointestinal disorders) | 3 | 0
Gastritis (Gastrointestinal disorders) | 3 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1
Oral pain (Gastrointestinal disorders) | 2 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Anal inflammation (Gastrointestinal disorders) | 1 | 0
Angular cheilitis (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 2
Glossitis (Gastrointestinal disorders) | 1 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 1 | 0
Lip swelling (Gastrointestinal disorders) | 1 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 1 | 0
Odynophagia (Gastrointestinal disorders) | 1 | 0
Oral dysaesthesia (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1
Gastric stenosis (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 15 | 4
Asthenia (General disorders) | 13 | 2
Pyrexia (General disorders) | 6 | 0
Oedema peripheral (General disorders) | 4 | 1
Mucosal inflammation (General disorders) | 2 | 0
Pain (General disorders) | 2 | 0
Chest discomfort (General disorders) | 1 | 0
Effusion (General disorders) | 1 | 0
Gait disturbance (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 1
Peripheral swelling (General disorders) | 1 | 0
Secretion discharge (General disorders) | 1 | 0
Tenderness (General disorders) | 1 | 0
Thirst (General disorders) | 1 | 0
Cholestasis (Hepatobiliary disorders) | 2 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 2 | 1
Hepatic cytolysis (Hepatobiliary disorders) | 1 | 0
Hepatic pain (Hepatobiliary disorders) | 1 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 0
Liver disorder (Hepatobiliary disorders) | 0 | 2
Paronychia (Infections and infestations) | 7 | 0
Urinary tract infection (Infections and infestations) | 7 | 0
Conjunctivitis (Infections and infestations) | 4 | 3
COVID-19 (Infections and infestations) | 2 | 0
Gingivitis (Infections and infestations) | 2 | 0
Abscess limb (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 1 | 1
Dermatophytosis of nail (Infections and infestations) | 1 | 0
Ear infection (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Onychomycosis (Infections and infestations) | 1 | 0
Oral candidiasis (Infections and infestations) | 1 | 0
Oral herpes (Infections and infestations) | 1 | 0
Oropharyngeal candidiasis (Infections and infestations) | 1 | 0
Otitis externa (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1
Tinea pedis (Infections and infestations) | 1 | 0
Tooth infection (Infections and infestations) | 1 | 0
Vaginal infection (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 3 | 0
Injury (Injury, poisoning and procedural complications) | 1 | 0
Neurological procedural complication (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 19 | 6
Aspartate aminotransferase increased (Investigations) | 15 | 7
Blood creatinine increased (Investigations) | 11 | 3
Gamma-glutamyltransferase increased (Investigations) | 6 | 1
Blood creatine phosphokinase increased (Investigations) | 5 | 0
Blood alkaline phosphatase increased (Investigations) | 4 | 2
Blood phosphorus increased (Investigations) | 4 | 0
Lymphocyte count decreased (Investigations) | 3 | 1
Weight decreased (Investigations) | 3 | 2
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0
Blood albumin abnormal (Investigations) | 1 | 0
Blood calcium increased (Investigations) | 1 | 0
Blood creatine increased (Investigations) | 1 | 0
Blood fibrinogen increased (Investigations) | 1 | 0
Blood magnesium decreased (Investigations) | 1 | 0
Blood thyroid stimulating hormone increased (Investigations) | 1 | 0
Blood triglycerides increased (Investigations) | 1 | 0
Blood urine present (Investigations) | 1 | 0
Creatinine renal clearance decreased (Investigations) | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0
Heart rate abnormal (Investigations) | 1 | 0
International normalised ratio increased (Investigations) | 1 | 0
Myoglobin blood increased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 1
Platelet count decreased (Investigations) | 1 | 0
SARS-CoV-2 test positive (Investigations) | 1 | 0
White blood cell count decreased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 2
Blood cholesterol increased (Investigations) | 0 | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 70 | 25
Decreased appetite (Metabolism and nutrition disorders) | 18 | 10
Hypercalcaemia (Metabolism and nutrition disorders) | 4 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 2
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 2
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 8 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Dysgeusia (Nervous system disorders) | 11 | 1
Headache (Nervous system disorders) | 5 | 2
Paraesthesia (Nervous system disorders) | 2 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 0
Ataxia (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0
Neuralgia (Nervous system disorders) | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 2 | 0
Depressed mood (Psychiatric disorders) | 1 | 0
Disorientation (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 2
Dysuria (Renal and urinary disorders) | 2 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Pyelocaliectasis (Renal and urinary disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 10 | 0
Onychomadesis (Skin and subcutaneous tissue disorders) | 7 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 6 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 4 | 1
Onycholysis (Skin and subcutaneous tissue disorders) | 4 | 0
Nail discolouration (Skin and subcutaneous tissue disorders) | 3 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 2 | 0
Eczema (Skin and subcutaneous tissue disorders) | 2 | 0
Nail dystrophy (Skin and subcutaneous tissue disorders) | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 1
Hair texture abnormal (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertrichosis (Skin and subcutaneous tissue disorders) | 1 | 0
Palmoplantar keratoderma (Skin and subcutaneous tissue disorders) | 1 | 0
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Embolism (Vascular disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
The Sponsor made a strategic decision to terminate the study considering enrollment challenges for some of the cohorts in the trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-12-10): https://cdn.clinicaltrials.gov/large-docs/45/NCT04189445/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-10): https://cdn.clinicaltrials.gov/large-docs/45/NCT04189445/SAP_001.pdf